CLINICAL TRIAL: NCT01027169
Title: An Open-label, Parallel-group, Single Centre, Single Oral Dose Study to Investigate the Pharmacokinetics of 50 mg Safinamide in Subjects With Mild and Moderate Hepatic Impairment as Compared to Matched Subjects With Normal Hepatic Function
Brief Title: A Study to Assess the Effect of Hepatic Impairment on Safinamide Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 28696
Record Dates: First submitted 2009-12-03; First posted 2009-12-07 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2011-08

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; Liver diseases; Pharmacokinetics; To Investigate Pharmacokinetics of Safinamide in Subjects With Mild and Moderate Hepatic Impairment as Compared to Healthy Subjects With Normal Hepatic Function
MeSH Terms: conditions — Liver Diseases | interventions — safinamide

ARMS (3):
- Arm 1 (Experimental): subjects with mild hepatic impairment
  Interventions: Drug: safinamide
- Arm 2 (Experimental): subjects with moderate hepatic impairment
  Interventions: Drug: safinamide
- Arm 3 (Experimental): matched subjects with normal hepatic function
  Interventions: Drug: safinamide

INTERVENTIONS:
Drug: safinamide — single dose of 50mg safinamide on Day 1
  Arms: Arm 1
Drug: safinamide — single dose of 50mg safinamide on Day 1
  Arms: Arm 2
Drug: safinamide — single dose of 50mg safinamide on Day 1
  Arms: Arm 3

SUMMARY:
The primary purpose of this study is to investigate the pharmacokinetics (behavior of the compound in the body) of safinamide in patients with different degrees of hepatic (liver) impairment in comparison to matched subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Hepatically impaired subjects - Subjects with liver cirrhosis and different degrees of impaired hepatic function: mild and moderate impaired hepatic function (Grade A, or B according to Child-Pugh classification)
* Healthy subjects - Subject is in good age-appropriate physical and mental health as established by medical history, physical examination, ECG and vital signs recordings, and results of biochemistry, haematology, coagulation and urinalysis testing within 3 weeks prior to the dosing
* All subject have given written informed consent before any study-related activities are carried out

Exclusion Criteria:

* Any clinically relevant disease or condition, which in the Investigator's opinion would exclude the subject from the study
* Diseases or surgeries of the gastrointestinal tract, which could influence the gastro-intestinal absorption and/or motility
* Hepatically impaired subjects - Subjects with primary biliary liver cirrhosis, hepatic encephalopathy grade III and IV, sepsis or spontaneous bacterial peritonitis, gastrointestinal bleeding within one month before the study, esophagus varices > grade II, acute hepatic failure of any aetiology, portosystemic shunt, renal impairment (creatinine clearance < 50 mL/min calculated by use of Cockroft Gault formula)
* Healthy subjects - Use of any medication, including multi-vitamin preparations, received within 21 days prior to the drug administration, or within six times the elimination half-life, whichever is longest, except combined oral contraceptives and occasional use of paracetamol or ibuprofen within 14 days before study drug administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of safinamide after single dose administration (Cmax) | 10 days
Pharmacokinetics of safinamide after single dose administration (AUC) | 10 days

SECONDARY OUTCOMES:
Safety and tolerability after single dose administration of safinamide (Adverse Events) | 12 days
Pharmacokinetics of safinamide metabolite NW1153 (Cmax) | 10 days
Pharmacokinetics of safinamide metabolite NW1153 (AUC) | 10 days
Pharmacokinetics of safinamide metabolite NW1689 (Cmax) | 10 days
Pharmacokinetics of safinamide metabolite NW1689 (AUC) | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Atef Halabi, MD, Principal Investigator — CRS Clinical Research Services Kiel GmbH
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany